CLINICAL TRIAL: NCT06802055
Title: Efficacy and Safety of Sirolimus With or Without Cyclosporin A in Chinese Patients With Aplastic Anemia Refractory/Intolerant to Cyclosporin A
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-25PJ0215
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Aplastic Anaemia
Keywords: Sirolimus; Relapsed/refractory aplastic anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Sirolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus + cyclosporin A (Experimental)
  Interventions: Drug: Sirolimus (Rapamune®); Drug: Cyclosporin A (CsA)
- Sirolimus (Placebo Comparator)
  Interventions: Drug: Sirolimus (Rapamune®)

INTERVENTIONS:
Drug: Sirolimus (Rapamune®) — Sirolimus 1-3 mg once daily orally, with a target trough blood concentration of 4-12 ng/ml.
Drug: Cyclosporin A (CsA) — Cyclosporine A 25-150 mg orally every 12 hours, with the dose adjusted based on renal function and trough concentration. For patients with normal renal function, the target trough concentration is approximately 150 ng/ml. For patients with impaired renal function, the cyclosporine A dose is reduced to 25-50 mg every 12 hours, aiming for recovery or stabilization of renal function.
  Arms: Sirolimus + cyclosporin A

SUMMARY:
This is a single center, randomized, open-label, phase II study to compare the efficacy of sirolimus combined with cyclosporin A (CsA) to sirolimus alone in Chinese subjects with aplastic anemia refractory/intolerant to CsA. The safety would also be evaluated. Patients would be randomized to receive sirolimus alone or sirolimus combined with CsA at a 1:3 ratio. Treatment with sirolimus will be started at 1-3 mg once daily orally, with a target trough blood concentration of 4-12 ng/ml. CsA will be given at 25-150 mg orally every 12 hours, with the dose adjusted based on renal function and trough concentration. For patients with normal renal function, the target trough concentration is approximately 150 ng/ml. For patients with impaired renal function, the cyclosporine A dose is reduced to 25-50 mg every 12 hours, aiming for recovery or stabilization of renal function. The hematological response rate and safety will be recorded and compared at 3 and 6 months after starting the study treatment (Week 13 and 25).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Diagnosed with acquired aplastic anemia (AA), excluding congenital AA;
3. At least one of the following criteria met at enrollment: hemoglobin < 100 g/L, platelets < 50 × 10⁹/L, or neutrophils < 1.0 × 10⁹/L;
4. At enrollment, meeting at least one of the following conditions:

   ① Cyclosporine A (CsA) ineffective: (CsA) used for at least 3 months without achieving partial response (PR), or disease relapse occurred;

   ② CsA intolerant: Unsuitable for standard dose CsA treatment due to adverse events or underlying conditions.
5. No active infections;
6. Not pregnant or breastfeeding;
7. Willing to sign the consent form;
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.

Exclusion Criteria:

1. Pancytopenia caused by other reasons, such as myelodysplastic syndrome (MDS);
2. Evidence of clonal hematopoietic system bone marrow diseases (e.g., MDS or acute myeloid leukemia, AML);
3. Paroxysmal nocturnal hemoglobinuria (PNH) clone ≥ 50%;
4. History of hematopoietic stem cell transplantation (HSCT) before enrollment;
5. Previous use of sirolimus or allergy to sirolimus;
6. Severe adverse events to CsA in the past, making it unsuitable for reuse;
7. Uncontrolled infection or bleeding with standard treatment;
8. Active infections with HIV, HCV, or HBV, liver cirrhosis, portal hypertension;
9. Any concurrent malignancy within the past 5 years, except for localized basal cell carcinoma of the skin;
10. History of thromboembolic events, myocardial infarction, or stroke (including antiphospholipid antibody syndrome), or current use of anticoagulants;
11. Pregnant or breastfeeding women;
12. Participation in other clinical trials within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) at 3 months | Week 12
  Overall Response Rate (ORR) is defined as the number of participants who meet the criteria of either complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Overall response rate (ORR) at 6 months | Week 24
  ORR will be evaluated after 6 months of treatment by measuring platelet, reticulocyte, hemoglobin, neutrophil and transfusion independence.
Changes in Hemoglobin in the Absence of Red Blood Cells Transfusion | Week 12
  The change in hematology values (hemoglobin) were evaluated
Changes in Platelet in the Absence of Platelet Transfusion | Week 12
  The change in hematology values (platelet) were evaluated
Duration of hematologic response | by 6 months (all patients), at 12 months (responders only)
  Time from the date of the start of the first response to the date of first relapse defined as again meeting criteria for aplastic anemia
Percentage of patients with clonal evolution to myelodysplasia, PNH, and acute leukemia | 12 months
  Clonal evolution to myelodysplasia is defined as a new marrow cytogenic abnormality with or without characteristic dysplastic marrow findings. Evolution to leukemia is defined as greater than 20% peripheral blood and/or marrow blasts. Evolution to paroxysmal nocturnal hemoglobinuria (PNH) is defined as a clone at baseline < 10% that rose to greater than 50% on study.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: Email request